CLINICAL TRIAL: NCT02376491
Title: Efficacy of Intermittent ThetaBurst Stimulation Compared to 10 Hz Stimulation on Dorsolateral Prefrontal Cortex in Treatment Resistant Major Depressive Disorder: a Double-blind Randomized Study
Acronym: THETA-DEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC14_0375
Record Dates: First submitted 2015-02-17; First posted 2015-03-03 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: DEPRESSION
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Frequency Left repetitive (Active Comparator): High Frequency Left repetitive transcranial magnetic stimulation five days per week for 4 weeks Magventure Cool B65 Coil with Magpro X100
  Interventions: Device: Transcranial magnetic stimulation
- intermittent Theta Burst Stimulation (iTBS) (Experimental): intermittent Theta Burst Stimulation (iTBS) five days per week for 4 weeks Magventure Cool B65 Coil with Magpro X100
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation

SUMMARY:
This trial will compare innovating stimulation parameters, intermittent Theta Burst Stimulation, to the standard high frequency stimulation protocol. The Left dorsolateral prefrontal cortex, targeted by MRI navigation will be the site of stimulation in both treatment conditions. The study seeks to determine if there is a superiority in therapeutic efficacy with iTBS protocol compared to conventional one.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 75 years
* Both gender eligible
* Volontary and able to give consent
* Major depressive episode (MADRS > 20) single or recurrent
* Resistance to at least 2 antidepressants ,
* Treated by antidepressant at efficient stable posology since more than 6 weeks

Exclusion Criteria:

* Initiation or modification of antidepressant drug
* Neurodegenerative diseas
* Bipolar I, II disorder
* Schizophrenia, schizoaffective disorder, schizophreniform, delusional disorder, or current psychotic symptoms
* Substance abuse in past 15 days
* Substance dependence not weaned
* Benzodiazepine and any anticonvulsant during rTMS treatment course
* ECT failure in medical history
* Contra-indication to rTMS and MRI
* Pregnancy
* Difficulty to obtain informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Therapeutic response rate | 6 months
  Primary outcome will be therapeutic response rate corresponding to with MADRS score improvement > 50 % in each group at the end of TMS sessions and one month after.
  A final score of <8 is categorized as remission.

SECONDARY OUTCOMES:
Relapse rate | 6 months
Quality of life | 6 months
Measures of cortical excitability | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Bulteau, dr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Derived] Bulteau S, Sebille V, Fayet G, Thomas-Ollivier V, Deschamps T, Bonnin-Rivalland A, Laforgue E, Pichot A, Valriviere P, Auffray-Calvier E, Fortin J, Pereon Y, Vanelle JM, Sauvaget A. Efficacy of intermittent Theta Burst Stimulation (iTBS) and 10-Hz high-frequency repetitive transcranial magnetic stimulation (rTMS) in treatment-resistant unipolar depression: study protocol for a randomised controlled trial. Trials. 2017 Jan 13;18(1):17. doi: 10.1186/s13063-016-1764-8. PMID 28086851